CLINICAL TRIAL: NCT01930630
Title: Extraesophageal Saline Injection Combined With EUS to Differentiate Between T3 and T4 Stage Esophageal Squamous Cell Carcinoma - A PhaseⅠTrial
Brief Title: ESI With EUS to Differentiate T3 and T4 ESCC
Acronym: ESI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian-jun Li, Associate Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ESI-2013; 2012-FXY-006 (Other: The ethic committee of Sun Yat-sen University Cancer Center)
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Esophageal Cancer
Keywords: extraesophageal saline injection (ESI);; esophageal squamous cell carcinoma (ESCC);; esophageal cancer;; endoscopic ultrasonography (EUS)
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extraesophageal saline injection (ESI) (Experimental): Extraesophageal saline injection (ESI) guided by EUS in patients with advanced ESCC preoperatively
  Interventions: Device: Extraesophageal saline injection (ESI)

INTERVENTIONS:
Device: Extraesophageal saline injection (ESI) — The patients with advanced ESCC are to undergo extraesophageal injection of 15ml saline preoperatively and subsequently detected by EUS to confirm whether saline separates esophagus from adjacent organs.
  Other Names: Extraesophageal saline injection;; Mucosal needle;; EUS:Fujinon7000(EG-530UR and EG-530UT)

SUMMARY:
By using a novel technique of extraesophageal saline injection (ESI),the esophagus is to be separate from the adjacent organs.The space between esophagus and adjacent organs can be detected by endoscopic ultrasonography enhanced with ESI.Therefore, ESI plus with EUS is to be differentiate between T3 and T4 stage esophageal squamous cell carcinoma (ESCC). The objective of this Phase Ⅰstudy is to confirm the safety and efficacy of ESI.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is one of the most common malignant tumors in the world, and China has the highest incidence of esophageal squamous cell carcinoma (ESCC).According to the TNM staging system of the Union for International Cancer Control (UICC) (7th Edition, 2012), EC invades the esophageal adventitia at the T3 stage; invades the pleura, pericardium and diaphragm at the T4a stage; and involves adjacent vital organs (mainly the thoracic aorta, aortic arch, trachea, tracheal bifurcation, and spine) at the T4b stage.It is considered that T3- and T4a-stage tumors can be surgically resected, while tumors at the T4b stage are not suitable for surgical resection.Therefore, it is important for physicians and patients to know whether the tumor has metastasized to adjacent organs before considering resection. The preoperative stage is unclear in many cases of progressive disease and the involvement of vital organs is only discovered by exploratory thoracotomy, because of which the resection may need to be terminated prematurely, leading to unnecessary injuries.Therefore, accurate preoperative staging of EC, especially during the later stages, is important for deciding the appropriate therapeutic option and evaluation of the prognosis.

The imaging methods used for preoperative staging of EC include endoscopic ultrasonography (EUS). However, EUS has poor accuracy in advanced ESCC, especially in T3 and T4 stage ESCC. Therefore, it is necessary to improve the preoperative accuracy of EUS for advanced EC.

Since extraesophageal space contains loose connective tissue and saline can permeate into extraesophageal space and separate esophagus from adjacent organ; furthermore, saline serves as an EUS contrast agent (negative) and is detected by EUS.Therefore, we envisaged that if saline is directly injected into extraesophageal space, the separation between the esophageal adventitia and its adjacent organs (especially the thoracic aorta, arcus aortae, and tracheal bifurcation) can be observed by EUS. In our recent experiment in canine model, guided by EUS,extraesophageal saline injection was successfully conducted and saline separated esophageal adventitia from adjacent organs including thoracic aorta, arcus aortae, trachea and bronchial bifurcation without any complication.

ELIGIBILITY:
Inclusion Criteria:

A)Age ranges 18-65 years old, no gander limited;

B)Patients with advanced ESCC (T2-T4) who were confirmed by standard endoscopy and pathologic biopsy;

C)Patients who agree to accept esophagectomy;

D)Patients with normal cardio-pulmonary and blood coagulation function; patients were predicted to be tolerated anesthesia and surgery;

E)Patients who understand the study, are willing to join this study and sign consent inform;

Exclusion Criteria:

1. Patients with early ESCC of Tis,T1a and T1b stages detected by standard EUS;
2. Patients cannot tolerate endoscopy and esophagectomy with various reasons;
3. Patients who have distant metastatic disease or multiple source of malignant tumor;
4. Patients with blood coagulation disorder;
5. Patients don't accept endoscopic or surgical resection subsequently;
6. Patients with poor compliancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 10 days
  Adverse events included bleeding due to great vessel split, asphyxia, esophageal perforation, acute heart failure or acute mediastinum inflammation during/post ESI.

SECONDARY OUTCOMES:
Efficacy of extraesophageal saline separating esophagus from adjacent organs detected by EUS or computerized tomography (CT) just after ESI | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Li, MD & PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China